CLINICAL TRIAL: NCT03803813
Title: The Incidence and Outcome of Sepsis After Craniocerebral Operation
Brief Title: Incidence of Sepsis After Craniocerebral Operation
Status: Completed | Type: Observational
Sponsor: Jianfang Zhou (Other)
Responsible Party: Sponsor-Investigator, Jianfang Zhou, Principal Investigator, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Other Study IDs: JZhou
Record Dates: First submitted 2018-12-26; First posted 2019-01-15 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Sepsis
Keywords: sepsis; septic shock; infection; craniotomy; outcome
MeSH Terms: conditions — Sepsis; Shock, Septic; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sepsis group: Patients have developed sepsis at ICU admission or during their ICU stay.
- non-sepsis group: Patients do not develope sepsis at ICU admission or during their ICU stay.

SUMMARY:
To investigate the incidence and outcome of sepsis in critical patients undergoing craniotomy.

DETAILED DESCRIPTION:
This is a prospective cohort study aiming to describe the incidence and outcome of sepsis in critical patients undergoing craniotomy. This study has been approved by the institutional review board of Beijing Tiantan hospital, and the need for informed consent was waived.

All patients over 18 years of age in intensive care will be screened for sepsis at admission or during their ICU stay, whereas those who stay in the ICU for <24 hrs for routine postoperative surveillance will be excluded. Patients readmitted into ICU and have been included at their first admission will not be included for a second time. Each center has one or more investigators who are residents of intensive care medicine and responsible for screening, patient records, and follow-up. They all have received at least one year of clinical training in critical care medicine and had previous research experience.

Sepsis and septic shock are diagnosed according to the sepsis 3.0 criteria. Acute organ dysfunction is defined as a Sequential Organ Failure Assessment (SOFA) score of 2 for the organ in question. The causal relationship between sepsis and organ dysfunction is confirmed based on medical recording and communication between the investigators and related ICU physicians. Infection is defined by the attending physicians as the presence of polymorphonuclear cells in a normally sterile body fluid(except blood),positive culture or Gram stain of a normally sterile body fluid or tissue, unquestionable clinical signs of infection, such as fecal peritonitis, necrotizing fasciitis, wound with purulent discharge, et al, or clinical suspected infection with corresponding antibiotic treatment. ICU-acquired infection is defined as infection identified 48 hours after ICU admission. Antibiotic consociation application is defined as the daily administration of more than one kind of the following antibiotics: penicillins, cephalosporins, carbapenem, macrolides, glycopeptides, aminoglycosides, quinolones, sulfonamides, and other antibiotics.

For patients developing sepsis at ICU admission or during their ICU stay, the following data will be collected using preprinted case report forms: age, sex, primary diagnosis, chronic comorbidities, clinical and laboratory data for admission Acute Physiology and Chronic Health Evaluation (APACHE) II and SOFA score, clinical and laboratory data for maximum SOFA score, microbiological and clinical infectious information, occurrence of ICU-acquired infection, antibiotics administered, hospital length of stay (LOS), ICU LOS, hospital costs, and outcome. For patients who have not developed severe sepsis at ICU admission or during the ICU stay, only age, sex, primary diagnosis, chronic comorbidities, ICU LOS, and outcome will be recorded. If a patient has more than one episode that meet the criteria, only the data from the first episode will be included in the study.

All recorded data will be screened in details by medical personnel for any missing information, logical errors, or insufficient details.

Continuous variables were expressed as mean (SD) and analyzed by unpaired Student's t test. Nonparametric variables were expressed as median and 25-75% percentiles and analyzed by the Mann-Whitney test. Categorical variables were expressed as absolute (n) and relative (%) frequency and were analyzed by chi-square test, as appropriate. p < 0.05 was considered statistically significant for all comparisons. SPSS version 19.0 for windows software was used for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* ICU length of stay ≥ 24 hours
* after craniotomy

Exclusion Criteria:

* <18 years
* ICU length of stay < 24 hours
* Patients or their immediate family members refuse to participate in the research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years of age and have undergone craniotomy in intensive care will be screened for sepsis at admission or during their ICU stay, whereas those who stay in the ICU for <24 hrs for routine postoperative surveillance will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 907 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of sepsis | 28 days
  The incidence of sepsis in critical patients undergoing craniotomy

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Study Chair — Beijing Tiantan Hospital, Capital Medical Universtity
Locations (1):
- Beijing Tian Tan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No